CLINICAL TRIAL: NCT06885268
Title: The Effect of Noradrenaline Infusion Versus Standard Blood Pressure Management on Perioperative HYPotension in NOn-caRdiac Surgery HYP-NOR Trial
Brief Title: Noradrenaline Versus Standard Blood Pressure Management for Perioperative Hypotension in Non-cardiac Surgery
Acronym: HYP-NOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Wojciech Szczeklik, Professor of Medical Sciences, Head of the Department of Intensive Care and Perioperative Medicine Faculty, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYP-NOR; 2023-508255-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure Management; Intraoperative Hypotension; Non-cardiac Surgery
Keywords: hypotension; noradrenaline infusion; perioperative care
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): In the intervention group, a standardized noradrenaline infusion at a concentration of 10 µg/mL will be initiated 15 to 60 seconds before induction of anaesthesia. The infusion will be titrated and maintained during surgery and postoperatively for up to 4 hours, with a minimum duration of 2 hours, until haemodynamic stability is achieved. Haemodynamic stability is defined as stable blood pressure requiring minimal noradrenaline support of 0.01 µg/kg/min or less for at least 1 hour. We will mandate avoidance of mean arterial pressure decreasing below 60 to 70 mm Hg. Once haemodynamic stability is achieved during the postoperative observation period, noradrenaline infusion may be discontinued. Safety criteria for discontinuation include systolic blood pressure above 180 mm Hg, in which case the infusion will be stopped. If systolic blood pressure is between 140 and 170 mm Hg, dose reduction or continuation at a very low noradrenaline infusion of 0.005 µg/kg/min, approximately 1 mL per h
  Interventions: Drug: noradrenaline infusion for management blood pressure
- Control group (Active Comparator): Standard blood pressure management reactive to blood pressure values. According to the 2022 ESA/ESC guidelines, patients in the control group will be treated to avoid a mean arterial pressure below 60 to 70 mm Hg. Ephedrine boluses (5 mg per bolus, up to a total intravenous dose of 25 mg) are recommended as first line treatment for hypotension. If hypotension persists, peripheral noradrenaline may be administered. Due to variability in clinical practice regarding the choice and timing of vasopressors and fluid therapy during and after surgery, further protocolization of hypotension management will not be mandated in order to enhance feasibility and generalizability of the trial.
  Interventions: Combination Product: standard blood pressure management

INTERVENTIONS:
Drug: noradrenaline infusion for management blood pressure — A single concentration of noradrenaline (10 μg/ml) will be initiated 15-60 seconds prior to the induction of anaesthesia, then titrated and maintained until 4 hours after surgery to meet pre-specified mean arterial pressure (MAP) targets. The drug infusion will be started at a dose of 0.01 μg/kg/min and will be titrated to a maximum of 0.1 μg/kg/min. Anaesthesiologists will be advised to use the lowest possible dose of noradrenaline. Avoidance of MAP decreases of >20% from baseline values or <60-70 mm Hg will be required in both groups. Individual baseline MAP value will be defined as resting blood pressure obtained in at least two measurements at the surgery ward on the day before surgery. Noradrenaline will be administered peripherally in all patients who do not have a central venous catheter in place.
  Arms: Intervention group
Combination Product: standard blood pressure management — Patients in the control group will receive standard blood pressure management reactive to blood pressure values. In the light of the current ESA/ESC 2022 guidelines, all patients in the control group will be treated to avoid MAP <60-70 mm Hg. Ephedrine boluses (5 mg each, up to 25 mg total intravenous dose) will be recommended as a first-line hypotension treatment. Subsequent treatment will involve administering peripheral noradrenaline. Notwithstanding, there is a variation in clinical practice regarding the choice and timing of vasopressors and fluids to be administered during and after surgery, therefore, hypotension treatment will not be further protocolized to increase the feasibility and generalizability of the trial.
  Arms: Control group

SUMMARY:
The effect of noradrenaline infusion versus standard blood pressure management on perioperative HYPotension in NOn-caRdiac surgery.

The study aims to determine whether perioperative noradrenaline infusion is superior to standard blood pressure management for the occurrence of perioperative hypotension.

DETAILED DESCRIPTION:
Patients will receive either noradrenaline infusion or standard blood pressure management during and up to 4 hours after surgery. Patients and health care providers will not be blinded to patients' allocation to either arm of the trial. Continuous blood pressure measurements will be secured in all patients who do not have an arterial line already in place for other indications using a non-invasive volume-clamp method. The medical team will not be aware of the continuous blood pressure monitoring and will use solely non-invasive blood pressure measurements at time intervals at least every 5 minutes in the operating room, and at least every 15 minutes in the post-anaesthesia care unit . In each group, patients will receive balanced crystalloids at 4 ml/kg per hour as maintenance fluid during surgery. In mechanical ventilation, a tidal volume of 8 mL/kg predicted body weight will be recommended. Other ventilatory settings, optimisation of volume status, depth of anaesthesia, patient positioning, as well as prompt diagnosis and treatment of reversible causes of hypotension will be prioritised in all patients in adherence with institutional protocols and current standards of practice.

The study aims to determine whether perioperative noradrenaline infusion can reduce exposure to hypotension compared to reactive treatment of hypotension, whether it is more effective in controlling hypotension during the intraoperatively and postoperatively, whether it reduces the risk of postoperative organ dysfunction, and whether it is safe and does not increase the risk of potential complications.

ELIGIBILITY:
Inclusion Criteria:

1. ≥45 years old
2. Elective or accelerated* non-cardiac surgery expected to last ≥1 hour and requiring general, neuraxial, or combined general with neuraxial anesthesia
3. Expected to stay overnight in the hospital after surgery
4. Written informed consent to participate in the HYP-NOR Trial provided
5. American Society of Anesthesiologists (ASA) physical status class II or higher.

Exclusion Criteria:

1. Newly diagnosed, untreated, or uncontrolled hypertension -in two measurements on the day before surgery Systolic Blood Pressure (SBP) ≥180 mm Hg or Diastolic Blood Pressure (DBP) ≥110 mm Hg
2. Persistent difference in recorded SBP between right and left upper limb >10 mm Hg
3. Persistent atrial fibrillation
4. Have a documented history of dementia
5. Have language, vision, or hearing impairments that may compromise cognitive assessments
6. Have a condition that precludes routine blood pressure management such as surgeon request for relative hypotension
7. Receiving irreversible nonselective monoamine oxidase inhibitors (e.g. tranylcypromine, phenelzine) within 2 weeks preceding study enrolment
8. The use of tricyclic antidepressants
9. Have Prinzmetal angina
10. Have contraindications to noradrenaline per clinician judgement
11. Noradrenaline infusion started before surgery or plan to use continuous noradrenaline infusion throughout the procedure
12. Treating physician (surgeon/anaesthetist) decides on the necessity of extended continuous hemodynamic monitoring during or after surgery
13. Severe kidney disease (MDRD creatinine clearance <15 mL/min/1.73m2) or renal replacement therapy
14. End-stage heart failure: defined as NYHA Class IV - severe limitations in daily activity. Patients experience symptoms even while at rest. Mostly bedbound patients.
15. Known severe liver disease: defined as the presence of liver cirrhosis or any of the symptoms of severe liver dysfunction: portal hypertension (esophageal varices, ascites), hepatocellular insufficiency (e.g., jaundice, hepatic encephalopathy) and coagulopathy (prolonged INR/APTT associated with known liver dysfunction).
16. Emergency and urgent surgery defined as performed within 24 hours of sudden illness/unplanned admission to hospital
17. Have previously participated in the trial: patient already took a part in the HYP-NOR trial in the past
18. Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative hypotension | During and up to 4 hours after surgery
  Number of episodes of perioperative hypotension defined as any mean arterial pressure (MAP) reading ≤55 mm Hg in the setting of a continuous blood pressure measurement.

SECONDARY OUTCOMES:
Myocardial Injury after Non-cardiac Surgery (MINS) | During hospitalization and up to 30 days after surgery
  Number of patients who experience MINS defined as any myocardial infarction and any acutely elevated postoperative cardiac troponin judged as resulting from myocardial ischemia using Roche's fifth generation Elecsys hsTnT, with an established cut-off of 20 ng/L combined with an absolute change of 5 ng/L or more (judged as due to ischemia)
Acute kidney injury fulfilling Kidney Disease Improving Global Outcomes (KDIGO) criteria | During hospitalization and up to 30 days after surgery
  Number of patients who experience an acute kidney injury (fulfilling KDIGO criteria)
Stroke | During hospitalization and up to 30 days after surgery
  Number of patients who experience a stroke is defined as a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting more than 24 hours or leading to death. Stroke will be sub-classified into hemorrhagic and non-hemorrhagic stroke.
Non-fatal cardiac arrest | During hospitalization and up to 30 days after surgery
  Number of patients who experience non-fatal cardiac arrest defined as successful resuscitation from either documented or presumed ventricular fibrillation, sustained ventricular tachycardia, asystole, or pulseless electrical activity (PEA) requiring cardiopulmonary resuscitation, pharmacological therapy, or cardiac defibrillation
Sepsis | During hospitalization and up to 30 days after surgery
  Number of patients who experience sepsis is defined as an increase in SOFA score of 2 or more, with evidence of infection. This outcome includes septic shock defined as sepsis with shock (vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mM [above18 mg/dL] in the absence of hypovolemia). Infection is defined as a pathologic process caused by the invasion of normally sterile tissue or fluid or body cavity by pathogenic or potentially pathogenic organisms.
Death | During hospitalization and up to 30 days after surgery
  Number of patients who die of any cause
Infusion-related reactions | During the infusion of noradrenaline and up to 30 days after drug administration, with assessment occurring postoperatively.
  The number of patients who experience infusion-related reactions, defined as disorders such as flushing, rash, fever, rigors, chills, dyspnoea, bronchospasms, cardiac dysfunction, and anaphylaxis. Grades of infusion site extravasation are defined according to the Common Terminology Criteria for Adverse Events.
Days alive and out of hospital | 30 days after surgery
  Number of days when a patient is alive and out of hospital
Clinically important atrial fibrillation | During hospitalization and up to 30 days after surgery
  Number of patients who experience clinically important atrial fibrillation, defined as new-onset atrial fibrillation or atrial flutter of any duration on an ECG or rhythm strip, which results in angina, congestive heart failure, symptomatic hypotension, or requires treatment with a rate-controlling drug, antiarrhythmic drug, or electrical cardioversion
Major bleeding | During hospitalization and up to 30 days after surgery
  Number of patients who experience an International Society on Thrombosis and Haemostasis (ISTH) major bleeding
Peripheral ischemia | During hospitalization and up to 30 days after surgery
  Number of patients who experience peripheral ischemia defined as the fingertip necrosis of upper and lower limbs

OTHER OUTCOMES:
Lowest MAP throughout the procedure | During surgery
  Number of patients who experience the lowest MAP throughout the procedure, defined as the lowest punctual measurement of mean arterial pressure
Median mean arterial pressure | During and up to 4 hours after surgery
Median heart rate | During and up to 4 hours after surgery
Acute Myocardial Infarction | During hospitalization and up to 30 days after surgery
  Number of patients who experience acute myocardial injury according to the Fourth Universal Definition of Myocardial Infarction as a detection of an elevated cTn value above the 99th percentile URL with a rise and/or fall of cTn values.
Peak troponin concentration | The first three days after surgery
  Peak troponin concentration
Area under the curve troponin | The first three days after surgery
  Area under the curve troponin is defined as total cTn release measured as area under the Troponin-Time curve
Bradycardia | During surgery, up to 4 hours after surgery, and up to 30 days after surgery.
  Number of patients who experience bradycardia, defined as a heart rate less than 40 beats per minute
Acute congestive heart failure | During hospitalization and up to 30 days after surgery
  Number of patients who experience acute congestive heart failure defined as an episode characterized by at least one of the following clinical signs (i.e. any of the following signs: elevated jugular venous pressure, respiratory rales/crackles, crepitations, or presence of S3) and at least one of the following: (I) Radiographic findings (i.e. vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema) OR (II) Heart failure treatment implemented with diuretics with documented clinical improvement
Acute Kidney Injury stage 2-3 | 30 days after surgery
  Number of patients who experience acute kidney injury stage 2-3 according to KDIGO criteria
Pneumonia | During hospitalization and up to 30 days after surgery
  Number of patients who experience pneumonia, defined according to the US Centers for Disease Control criteria
Postoperative pulmonary complications | During hospitalization and up to 30 days after surgery
  Number of patients who experience postoperative pulmonary complications which are a composite outcome comprised of the following outcomes: 1. Atelectasis detected on computed tomography or chest radiograph 2. Pneumonia using US Centers for Disease Control criteria 3. Acute respiratory distress syndrome (according to Berlin definition) 4. Pulmonary aspiration (clear clinical history AND radiological evidence)
Surgical site infection | During hospitalization and up to 30 days after surgery
  Number of patients who experience surgical site infection defined according to the Centers for Disease Control and Prevention (CDC) criteria
Postoperative delirium | Assessment on postoperative days 1, 2, 3
  Number of patients who experience delirium (based on The Nursing Delirium Screening Scale - NuDESC). A total score of 2 or higher on the scale indicates a positive result for the diagnosis of delirium.
Discharge destination | 30 days after surgery
  Number of patients discharged from the hospital to home/long-term care facility/other
Cognitive decline | 30 days after surgery
  Number of patients who experience cognitive decline (defined as a decline of at least 2 points on the Montreal Cognitive Assessment, MoCA, performed via telephone) compared to the assessment conducted after consent and before randomization
Days alive and outside the intensive care unit | 30 days after surgery
  Number of days when a patient is alive and outside the intensive care unit
Health-related quality of life | 30 days after surgery
  Health-related quality of life will be evaluated (based on the EuroQol 5 Dimension, five-level version [EQ-5D]), compared to the assessment made after consent and before randomization.
Lowest MAP during the 4 hours postoperative period | up to 4 hours after surgery
  The lowest recorded mean arterial pressure during postoperative monitoring lasting at least 2 hours and up to 4 hours after surgery.
Perioperative myocardial infarction/injury | up to 72 hours (3 days) postoperatively
  Number of Participants with Perioperative myocardial infarction/injury as defined by the 2022 European Society of Cardiology (ESC) Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery: an absolute increase in hs-cTn concentration of more than the 99th percentile URL after surgery compared to the pre-operative level. In the absence of a preoperative hs-cTn T/I concentration, a hs-cTn more than five-times the 99th percentile URL or an absolute increase or decrease more than the 99th percentile URL

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Szczeklik, MD, PhD, Study Director — Centre for Intensive Care and Perioperative Medicine, Jagiellonian University Medical College
Locations (5):
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne im. Prof. Kornela Gibińskiego Śląski Uniwersytet Medyczny, Katowice
  - 5 Wojskowy Szpital Kliniczny z Polikliniką Samodzielny Publiczny Zakład Opieki Zdrowotnej w Krakowie, Krakow
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, Zabrze

IPD SHARING:
Plan to Share IPD: No